CLINICAL TRIAL: NCT02806531
Title: Safety Study of Enterovirus 71 Vaccine in Children Aged 6-35 Months Old
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Chaoyang District Centre for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: cycdc2016-2
Record Dates: First submitted 2016-06-16; First posted 2016-06-20 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Enterovirus 71 Vaccine
Keywords: vaccine; safety

ARMS (1):
- two doses enterovirus 71 vaccine (Experimental): Two doses of enterovirus 71 vaccine will be given in aged 6-35 months old, 28 days interval.
  Interventions: Biological: two doses enterovirus 71 vaccine

INTERVENTIONS:
Biological: two doses enterovirus 71 vaccine — Two doses of enterovirus 71 vaccine will be given in children aged 6-35 months old, 28 days interval.

SUMMARY:
This phase IV clinical study evaluates the safety of enterovirus 71 vaccine in children aged 6-35 months old by the method of both passive and active surveillance.

ELIGIBILITY:
Inclusion Criteria:

* Infant and toddlers aged 6 and 35 months, meeting the criteria of receiving vaccine based on the judgement of caregivers at vaccination clinic. And The legal guardian are willing to vaccination at his own expense.

Exclusion Criteria:

* History of allergy to any vaccine ingredient or gentamycin;
* Fever, or acute disease, or acute stage of chronic disease;
* Having serious chronic diseases, or allergic constitution;
* Refusal of follow-up for safety concern.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20000 (Estimated)
Dates: Start 2016-07; Primary Completion 2018-07 (Estimated)

PRIMARY OUTCOMES:
The rate of adverse reactions of enterovirus 71 Vaccine | 28 days
  Adverse reactions associated with vaccine will be observed in subjects after each vaccination. Solicited local adverse events include Pain, Redness, Swelling, Induration, Rash, Pruritus at injection site. solicited general adverse events include Fever, Nausea, Vomiting, Diarrhea, Decreased appetite, Be agitated (irritability, abnormal crying), fatigue, allergy